CLINICAL TRIAL: NCT01920555
Title: Double-Blind, Placebo-Controlled Trial of Ketamine Therapy in Treatment-Resistant Depression (TRD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Baylor College of Medicine (Other); Icahn School of Medicine at Mount Sinai (Other); Stanford University (Other); University of Texas (Other); Yale University (Other)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Overall Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAP-003; 271201100006I-0-27100007-1 (NIH)
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Treatment Resistant Depression
Keywords: Depression; Treatment Resistant Depression; Ketamine; Antidepressant; MDD; Major Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Ketamine 0.1mg (Active Comparator): Patients in this arm will receive 0.1 mg/kg of Ketamine - one single infusion
  Interventions: Drug: Ketamine
- Ketamine 0.2mg (Active Comparator): Patients in this arm will receive 0.2 mg/kg of Ketamine - one single infusion
  Interventions: Drug: Ketamine
- Ketamine 0.5mg (Active Comparator): Patients in this arm will receive 0.5 mg/kg of Ketamine - one single infusion
  Interventions: Drug: Ketamine
- Ketamine 1.0mg (Active Comparator): Patients in this arm will receive 1.0 mg/kg of Ketamine - one single infusion
  Interventions: Drug: Ketamine
- Midazolam (Active Placebo) (Placebo Comparator): Patients in this arm will receive 0.045 mg/kg of midazolam - one single infusion
  Interventions: Drug: Placebo Midazolam

INTERVENTIONS:
Drug: Ketamine — Dose of Ketamine will be 0.1 mg/kg - one single infusion
  Arms: Ketamine 0.1mg
Drug: Ketamine — Dose of Ketamine will be 0.2 mg/kg - one single infusion
  Arms: Ketamine 0.2mg
Drug: Ketamine — Dose of Ketamine will be 0.5 mg/kg - one single infusion
  Arms: Ketamine 0.5mg
Drug: Ketamine — Dose of Ketamine will be 1.0 mg/kg - one single infusion
  Arms: Ketamine 1.0mg
Drug: Placebo Midazolam — Dose of Midazolam (active placebo) will be 0.045 mg/kg - one single infusion
  Arms: Midazolam (Active Placebo)

SUMMARY:
This study is looking at the efficacy, durability, safety, and tolerability of multiple single doses of Ketamine vs. active placebo for treating patients with treatment resistant depression who are taking an antidepressant that is not working for them.

DETAILED DESCRIPTION:
The primary objective is to investigate whether all doses (0.1 mg/kg, 0.2 mg/kg, 0.5 mg/kg, and 1.0 mg/kg) of ketamine are superior to active placebo (midazolam 0.045 mg/kg) therapy in the acute treatment of patients with treatment resistant depression within 72 hours (Day 3), when added to ongoing and stable antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-70 years old.
* Able to read, understand, and provide written, dated informed consent prior to screening.
* Diagnosed with Major Depressive Disorder (MDD), single or recurrent, and currently experiencing a Major Depressive Episode (MDE) of at least eight weeks in duration, prior to screening.
* Has a history of TRD during the current MDE.
* Meet the threshold on the total MADRS score of greater than or equal to 20 at both screening and baseline visits (Day -7/-28 and Day 0), as confirmed by the remote centralized MGH CTNI rater between the screen visit and the baseline visit.
* In good general health
* For female participants, status of non-childbearing potential or use of an acceptable form of birth control
* Body mass index between 18-35 kg/m2
* Concurrent psychotherapy will be allowed if the type and frequency of the therapy has been stable for at least three months prior to screening and is expected to remain stable during participation in the study
* Concurrent hypnotic therapy will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

Exclusion Criteria:

* Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study
* Female that is pregnant or breastfeeding
* Female with a positive pregnancy test at screening or baseline
* History during the current MDE of failure to achieve a satisfactory response to >7 treatment courses of a therapeutic dose of an antidepressant therapy of at least 8 weeks duration during the current episode
* Total MADRS score of <20 at the screen or baseline visits, or as assessed by the remote, independent MGH CTNI rater and reported to the site
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence) with the exception of nicotine dependence, at screening or within 6 months prior to screening
* Current Axis I disorder that is the principal focus of treatment and MDD the secondary focus of treatment for the past 6 months or more
* History of bipolar disorder, schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes
* History of eating disorders within five years of screening
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant at any time within 6 months prior to screening
* Subject is considered at significant risk for suicidal behavior during the course of their participation in the study
* Has failed to respond to electroconvulsive therapy (ECT) during the current depressive episode
* Has received vagus nerve stimulation (VNS) at any time prior to screening
* Has dementia, delirium, amnestic, or any other cognitive disorder
* Has a clinically significant abnormality on the screening physical examination
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation
* Current episode of:

  1. Hypertension, Stage 1 as defined by a systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90 mmHg at screening on two of three measurements (standing and supine) at least 15 minutes apart.
  2. Hypertension, Stage 1 as defined by a systolic blood pressure ≥155 mmHg or diastolic blood pressure ≥99 mmHg at the Baseline Visit (Visit 1) within 1.5 hours prior to randomization on two of three measurements (standing and supine) at least 15 minutes apart.
  3. Recent myocardial infarction (within one year) or a history of myocardial infarction.
  4. Syncopal event within the past year.
  5. Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2
  6. Angina pectoris.
  7. Heart rate <50 or >105 beats per minute at screening or randomization (Baseline Visit).
  8. QTcF (Fridericia-corrected) ≥450 msec at screening or randomization (Baseline Visit).
* Current history of hypertension, or on antihypertensives for the purpose of lowering blood pressure, who have either had an increase in antihypertensive dose or increase in the number of antihypertensive drugs used to treat hypertension over the last 2 months.
* Chronic lung disease excluding asthma.
* Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system disorder, epilepsy, mental retardation, or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system, or a history of significant head trauma within the past 2 years
* Presents with any of the following lab abnormalities:

  1. Thyroid stimulating hormone outside of the normal limits and clinically significant as determined by the investigator. Free thyroxine (T4) levels may be measured if TSH level is high. Subject will be excluded if T4 level is clinically significant.
  2. Patients with diabetes mellitus fulfilling any of the following criteria:

  i. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.5% at screening ii. Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus related illness in the past 12 weeks iii. Not under physician care for diabetes mellitus iv. Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.

  c. Any other clinically significant abnormal laboratory result (as determined after evaluation by study investigator and MGH CTNI medical monitor) at the time of the screening exam.
* History of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than 2 months prior to screening. (Subjects on a stable dosage of thyroid replacement medication for at least 2 months or more prior to screening are eligible for enrollment.)
* History of hyperthyroidism which was treated (medically or surgically) less than six months prior to screening
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation
* History of positive screening urine test for drugs of abuse at screening
* Patients with exclusionary laboratory values, or requiring treatment with exclusionary concomitant medications
* Patients on exclusionary concomitant psychotropic medications, the half-life of which would not allow sufficient time for patients to have been free of the medication post-taper for five half-lives within the maximum screening period (28 days).
* Patient who have participated in studies of ketamine or AZD6765 or other NMDA receptor antagonists for depression and received active treatment.
* Patients with narrow angle glaucoma
* Patients with a lifetime history of PCP/Ketamine drug use
* Liver Function Tests higher than 2.5 times upper limit of normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Guy W, editor. ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: US Department of Heath, Education, and Welfare Public Health Service Alcohol, Drug Abuse, and Mental Health Administration; 1976.
- [Background] Nierenberg AA, Bentley KH, Farabaugh AH, Fava M, Deckersbach T. The absence of depressive symptoms is not the presence of wellness: validation of the Clinical Positive Affect Scale. Aust N Z J Psychiatry. 2012 Dec;46(12):1165-72. doi: 10.1177/0004867412459810. Epub 2012 Sep 18. PMID 22990434
- [Background] Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007 Jul;164(7):1035-43. doi: 10.1176/ajp.2007.164.7.1035. PMID 17606655
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Bremner JD, Krystal JH, Putnam FW, Southwick SM, Marmar C, Charney DS, Mazure CM. Measurement of dissociative states with the Clinician-Administered Dissociative States Scale (CADSS). J Trauma Stress. 1998 Jan;11(1):125-36. doi: 10.1023/A:1024465317902. PMID 9479681
- [Derived] Feeney A, Hoeppner BB, Freeman MP, Flynn M, Iosifescu DV, Trivedi MH, Sanacora G, Mathew SJ, DeBattista C, Ionescu DF, Cusin C, Papakostas GI, Jha MK, Fava M. Effect of Concomitant Benzodiazepines on the Antidepressant Effects of Ketamine: Findings From the RAPID Intravenous Ketamine Study. J Clin Psychiatry. 2022 Nov 14;84(1):22m14491. doi: 10.4088/JCP.22m14491. PMID 36383742
- [Derived] Feeney A, Hock RS, Freeman MP, Flynn M, Hoeppner B, Iosifescu DV, Trivedi MH, Sanacora G, Mathew SJ, Debattista C, Ionescu DF, Fava M, Papakostas GI. The effect of single administration of intravenous ketamine augmentation on suicidal ideation in treatment-resistant unipolar depression: Results from a randomized double-blind study. Eur Neuropsychopharmacol. 2021 Aug;49:122-132. doi: 10.1016/j.euroneuro.2021.04.024. Epub 2021 Jun 3. PMID 34090255
- [Derived] Freeman MP, Hock RS, Papakostas GI, Judge H, Cusin C, Mathew SJ, Sanacora G, Iosifescu DV, DeBattista C, Trivedi MH, Fava M. Body Mass Index as a Moderator of Treatment Response to Ketamine for Major Depressive Disorder. J Clin Psychopharmacol. 2020 May/Jun;40(3):287-292. doi: 10.1097/JCP.0000000000001209. PMID 32332464
- [Derived] Fava M, Freeman MP, Flynn M, Judge H, Hoeppner BB, Cusin C, Ionescu DF, Mathew SJ, Chang LC, Iosifescu DV, Murrough J, Debattista C, Schatzberg AF, Trivedi MH, Jha MK, Sanacora G, Wilkinson ST, Papakostas GI. Double-blind, placebo-controlled, dose-ranging trial of intravenous ketamine as adjunctive therapy in treatment-resistant depression (TRD). Mol Psychiatry. 2020 Jul;25(7):1592-1603. doi: 10.1038/s41380-018-0256-5. Epub 2018 Oct 3. PMID 30283029

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening period served as a wash-out period for any prohibited medications that could be discontinued safely. Discontinuation of medications were discussed in consultation with the prescribing clinician.
Period: Overall Study
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam (Active Placebo)
Started | 18 | 20 | 22 | 20 | 19
Completed | 14 | 16 | 21 | 17 | 18
Not Completed | 4 | 4 | 1 | 3 | 1
Not completed — Physician Decision | 1 | 2 | 1 | 2 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Travel Difficulties | 1 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam (Active Placebo) | Total
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.9) | 45.5 (14.6) | 48.6 (12.9) | 47.4 (10.1) | 45.6 (13.8) | 46.04 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 11 | 8 | 11 | 49
  Male | 8 | 11 | 11 | 12 | 8 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 17 | 20 | 20 | 20 | 19 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (3.1) | 24.9 (3.7) | 25.3 (5.7) | 26.1 (3.8) | 26.3 (4.1) | 24.96 (4.08)
Abnormal and Clinically Significant Labs [Count of Participants; unit: Participants] — Collected at Screening and Day 0 (Day 0 is pre-treatment) CBC, Chemistry (Total bilirubin, AST, ALT, GGT, ALK Phosphatase, Creatinine, BUN/Urea, Glucose, Uric Acid),Hormonal Measures in female subjects: Estradiol, Progesterone, FSH, LH, SHBG, Testosterone; Free testosterone, Hormonal Measures in male subjects: Testosterone, free testosterone, SHBG, DHEA, Progesterone, TSH, Pregnancy Test, Urine Tox Screen
  Participants
    CBC | 0 | 0 | 0 | 0 | 0 | 0
    Chemistry | 0 | 0 | 0 | 0 | 0 | 0
    Hormonal Measures (testosterone, SHBG, Free T) | 0 | 2 | 0 | 0 | 0 | 2
    Hormonal Measures (DHEA) | 0 | 0 | 0 | 1 | 0 | 1
    Hormonal Measures (remaining tests) | 0 | 0 | 0 | 0 | 0 | 0
    Pregnancy Test | 0 | 0 | 0 | 0 | 0 | 0
    Urine Toxicology Screen | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression - 6 Items
Description: The HAMD6 is a 6-item clinician-rated scale, where clinicians rate the presence of depression symptoms (i.e., depressed mood, guilt, work and interests, psychomotor retardation, psychic anxiety, somatic symptoms) on a 5-point scale, where 0 = not present, and 1-4 represent increasingly severe symptoms. One item (i.e., somatic symptoms) is rated on only a 3-point scale, ranging from 0-2. The possible scale range is 0-22, where higher values represent more severe depression. This instrument is completed with a structured interview guide by the clinician based on his/her assessment of the patient's symptoms. This structured interview has been validated for use with time frames shorter than one week. In this study, the HAMD6 was used to assess symptoms occurring in the past 24 hours.
Time Frame: A baseline assessment was made on Day 0, preceding infusion (i.e., treatment). Outcome assessments were made on days 1, 3, 5, 7, 14, and 30. The primary endpoint for this study was Day 3. Thus, the outcome measure table provides data on Days 0, 1, & 3
Population: Several subjects dropped out of the study in between Day 0, Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Midazolam 0.045mg: Patients in this arm will receive 0.045 mg/kg of Midazolam (active placebo) - one single infusion
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Day 0 | 12.5555556 (1.8221585) | 12.7500000 (2.4894514) | 12.5909091 (1.4690162) | 12.6315789 (2.0872770) | 13.0526316 (2.2967050)
  Day 1: number analyzed (Participants) | 16 | 20 | 22 | 20 | 19
  Day 1 | 7.5000000 (4.3204938) | 9.2631579 (3.6944719) | 5.8636364 (4.4859087) | 6.9000000 (4.5061362) | 10.6666667 (3.3606722)
  Day 3: number analyzed (Participants) | 15 | 19 | 22 | 20 | 19
  Day 3 | 6.8000000 (4.6167397) | 8.4736842 (4.9818384) | 5.9047619 (4.3000554) | 7.2000000 (3.8196170) | 9.0555556 (4.5435439)
Statistical Analysis 1: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.1mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.14, Mixed Models Analysis — Holm's method was applied to the model-produced differences of least squares for the eight a priori identified contrasts of interest, that is, the difference between each ketamine group vs. placebo at Days 1 and 3; Mean Difference (Final Values) = -3.18, 95% CI 2-sided [-5.93 to -0.43]
Statistical Analysis 2: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.2mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.79, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-3.75 to 1.49]
Statistical Analysis 3: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.5mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.79, 95% CI 2-sided [-7.35 to -2.24]
Statistical Analysis 4: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 1.0mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.04, Mixed Models Analysis; Mean Difference (Final Values) = -3.76, 95% CI 2-sided [-6.37 to -1.15]
Statistical Analysis 5: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.1mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.72, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-5.04 to 0.95]
Statistical Analysis 6: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.2mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.80, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-3.18 to 2.46]
Statistical Analysis 7: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.5mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.14, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.12, 95% CI 2-sided [-5.97 to -0.44]
Statistical Analysis 8: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 1.0mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.72, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-4.65 to 0.96]

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item clinician-rated scale measuring depression severity. Symptoms are rated on a 7-point scale, where 0 = "not present", and 1-6 represent increasing severity. Values 2, 4, and 6 have specific anchoring text (e.g., 2="Difficulties in starting activities." 4="Difficulties in starting simple routine activities which are carried out with effort, 6="Complete lassitude. Unable to do anything without help.") Values 1, 3, and 5 do not have specific text. The possible scale range is 0-60, where higher values represent higher severity. In this study, the MADRS was used to rate symptoms occurring in the past 3 days.
Time Frame: A baseline assessment was made on Day 0, preceding infusion (i.e., treatment). Outcome assessments were made on days 3, 5, 7, 14, and 30. The primary endpoint for this study was Day 3. Thus, the outcome measure table provides data on Days 0 and 3.
Population: Several subjects dropped out of the study in between Day 0, Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Day 0 | 33.8333333 (5.9334545) | 34.4500000 (8.4571676) | 31.5909091 (3.9359042) | 32.6500000 (5.8873191) | 33.6315789 (7.0884141)
  Day 3: number analyzed (Participants) | 15 | 19 | 21 | 20 | 18
  Day 3 | 19.6666667 (10.8144524) | 22.6315789 (11.7294052) | 14.7619048 (8.9883523) | 17.1000000 (11.5708345) | 24.8333333 (10.5286723)
Statistical Analysis 1: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.1 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were four pairwise comparisons of interest (see Analysis 1-4), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.33, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.15, 95% CI 2-sided [-12.44 to 2.14]
Statistical Analysis 2: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.2 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were four pairwise comparisons of interest (see Analysis 1-4), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.53, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-9.03 to 4.72]
Statistical Analysis 3: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.5 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were four pairwise comparisons of interest (see Analysis 1-4), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.85, 95% CI 2-sided [-16.56 to -3.15]
Statistical Analysis 4: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 1.0 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were four pairwise comparisons of interest (see Analysis 1-4), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.72, 95% CI 2-sided [-14.52 to -0.93]

3. Secondary Outcome: Clinical Global Impressions-Severity (CGI-S)
Description: The CGI-S is a clinician rated single-item scale: "How depressed is the patient at this time?", rated on a 7-point response scale: 1 = Normal, not at all depressed, 2 = Borderline depressed, 3 = Mildly depressed, 4 = Moderately depressed. 5 = Markedly depressed, 6 = severely depressed, 7 = Among the most severely depressed patients. When rating patients, clinicians were asked to consider the past 24 hours.
Time Frame: A baseline assessment was made on Day 0, preceding infusion (i.e., treatment). Outcome assessments were made on days 1, 3, 5, 7, 14, and 30. The primary endpoint for this study was Day 3. Thus, the outcome measure table provides data on Days 0, 1 and 3
Population: Several subjects dropped out of the study in between Day 0, Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Day 0 | 5.0000000 (0.7669650) | 5.2000000 (0.6958524) | 4.8636364 (0.6396021) | 5.2000000 (0.7677719) | 5.000000 (0.7453560)
  Day 1: number analyzed (Participants) | 16 | 19 | 22 | 20 | 18
  Day 1 | 3.5625000 (1.4591664) | 4.2631579 (1.2401660) | 3.2727273 (1.2792043) | 3.5000000 (1.1002392) | 4.555556 (0.7838234)
  Day 3: number analyzed (Participants) | 15 | 19 | 21 | 20 | 18
  Day 3 | 3.4000000 (1.6388149) | 3.7368421 (1.4848159) | 3.1428571 (1.3887301) | 3.3000000 (1.4545754) | 4.1666667 (1.3394468)
Statistical Analysis 1: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.1 mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-1.83 to -0.22]
Statistical Analysis 2: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.2 mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.82, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.02 to 0.51]
Statistical Analysis 3: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.5 mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.00720, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.02 to -0.54]
Statistical Analysis 4: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 1.0 mg/kg vs. midazolam at Day 1: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.04884, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.81 to -0.29]
Statistical Analysis 5: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.1 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.48, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.70 to 0.28]
Statistical Analysis 6: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.2 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.82, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.32 to 0.55]
Statistical Analysis 7: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 0.5 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.16, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.91 to -0.09]
Statistical Analysis 8: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; Ketamine 1.0 mg/kg vs. midazolam at Day 3: As estimated by the repeated measures fixed effects model with DAY (0, 1, 3), GROUP (5 groups as specified above), and the DAY*GROUP interaction effect. Because there were eight pairwise comparisons of interest (see Analysis 1-8), we used Holm's method to protect family-wise error rate in the presence of multiple testing; Test type: Superiority; p = 0.27, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.78 to 0.07]

4. Secondary Outcome: Clinical Global Impressions-Improvement (CGI-I) Scale
Description: The CGI-I is a clinician rated single-item scale: "Compared to the patient's condition at admission, how much has the patient changed?", rated on a 7-point response scale: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, and 7 = Very much worse. In this case, "admission" referred to the CGI-S screening assessments performed between Day -28 an -7, one conducted during the screening visit, and a second rating conducted by a remote, independent rater.
Time Frame: as for outcome 3
Population: Several subjects dropped out of the study in between Day 0, Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Day 0 | 3.8888889 (0.3233808) | 4.0500000 (0.2236068) | 4.1363636 (0.7101613) | 4.0000000 (0.4588315) | 4.1578947 (0.6021404)
  Day 1: number analyzed (Participants) | 16 | 19 | 22 | 20 | 18
  Day 1 | 3.0625000 (1.4361407) | 3.3684211 (1.0651305) | 2.6363636 (0.9021379) | 3.0500000 (1.2343760) | 3.6111111 (0.6076850)
  Day 3: number analyzed (Participants) | 15 | 19 | 22 | 20 | 18
  Day 3 | 2.9333333 (1.2798809) | 2.8421053 (1.2588865) | 2.5714286 (0.9258201) | 2.5500000 (1.0990426) | 3.1666667 (1.0431852)
Statistical Analysis 1: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.54, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.54, 95% CI 2-sided [-1.25 to 0.17]
Statistical Analysis 2: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.78 to 0.58]
Statistical Analysis 3: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-1.64 to -0.31]
Statistical Analysis 4: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.54, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.24 to 0.11]
Statistical Analysis 5: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.96 to 0.57]
Statistical Analysis 6: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.93 to 0.51]
Statistical Analysis 7: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.52, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.35 to 0.06]
Statistical Analysis 8: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p = 0.54, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.33 to 0.10]

5. Secondary Outcome: Symptoms of Depression Questionnaire (SDQ)
Description: The SDQ is a 44-item self-report scale, which aims to measure depression more comprehensively by including the assessment of symptoms in the anxiety-depression spectrum, including symptoms of irritability, anger attacks, and anxiety. Items are rated on an 6-point Likert scale, where participants are asked to rate if a specific symptom (e.g. "How has your mood been over the past 24 hours?") is normal for him or her (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). The total scale score is calculated by averaging across the items, resulting in a possible range from 1 to 6. Higher scores indicate greater depression severity. When rating, patients were asked to consider their symptoms during the past 24 hours.
Time Frame: as for outcome 3
Population: Several subjects dropped out of the study in between Day 0, Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Day 0 | 3.5164141 (0.5081856) | 3.4636364 (0.5416735) | 3.5392562 (0.5838397) | 3.4113636 (0.4336652) | 3.4264507 (0.4719770)
  Day 1: number analyzed (Participants) | 16 | 19 | 22 | 20 | 18
  Day 1 | 2.5752843 (0.7091841) | 2.9096195 (0.7123910) | 2.3109504 (0.6315677) | 2.6113636 (0.500567) | 2.9200573 (0.6464210)
  Day 3: number analyzed (Participants) | 15 | 18 | 21 | 20 | 18
  Day 3 | 2.5106061 (0.7158120) | 2.7828283 (0.7398734) | 2.5573593 (0.9017779) | 2.5909091 (0.5736341) | 2.8751353 (0.6668931)
Statistical Analysis 1: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.74, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.79 to 0.08]
Statistical Analysis 2: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.37 to 0.45]
Statistical Analysis 3: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.02, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.01 to -0.21]
Statistical Analysis 4: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.80, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.72 to 0.10]
Statistical Analysis 5: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.88, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.83 to 0.18]
Statistical Analysis 6: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.53 to 0.44]
Statistical Analysis 7: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.88, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.79 to 0.15]
Statistical Analysis 8: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p = 0.88, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.76 to 0.19]

6. Secondary Outcome: Clinical Positive Affect Scale (CPAS)
Description: The CPAS is a 16-item self-report scale to assess the level to which participants experience persistent distress due to feeling that they have not returned to their normal or premorbid state. Items (e.g., "I look forward to things") are rated on a 5-point scale (0=not at all, 1=very much less than normal, 2=much less than normal, 3=slightly less than normal, 4=same as best or normal self). The possible scale range is 0 to 64, with higher scores indicating greater recovery from depression. Patients were asked to rate their experience of the past 24 hours.
Time Frame: as for outcome 3
Population: Several subjects dropped out of the study in between Day 0, Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Day 0 | 19.3333333 (12.1896774) | 20.5000000 (15.4357753) | 20.6363636 (11.7008158) | 21.2500000 (14.6785737) | 21.2631579 (12.1052886)
  Day 1: number analyzed (Participants) | 16 | 19 | 22 | 20 | 18
  Day 1 | 35.2500000 (20.9936498) | 27.0526316 (18.8516833) | 40.8696964 (19.5284785) | 33.0000000 (16.2642650) | 24.4444444 (15.2053482)
  Day 3: number analyzed (Participants) | 15 | 18 | 21 | 20 | 16
  Day 3 | 38.8666667 (22.8666667) | 28.3888889 (20.2459550) | 39.7619048 (22.5319878) | 37.4500000 (18.7096232) | 33.3750000 (15.8445574)
Statistical Analysis 1: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.49, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.18, 95% CI 2-sided [-0.94 to 23.29]
Statistical Analysis 2: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.37, 95% CI 2-sided [-10.19 to 12.93]
Statistical Analysis 3: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.03, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 16.54, 95% CI 2-sided [5.31 to 27.77]
Statistical Analysis 4: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.82, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.68, 95% CI 2-sided [-2.81 to 20.16]
Statistical Analysis 5: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.11, 95% CI 2-sided [-8.83 to 19.05]
Statistical Analysis 6: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.64, 95% CI 2-sided [-19.87 to 6.59]
Statistical Analysis 7: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.64, 95% CI 2-sided [-5.26 to 20.53]
Statistical Analysis 8: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.80, 95% CI 2-sided [-8.31 to 17.91]

7. Secondary Outcome: Snaith-Hamilton Pleasure-Scale (SHAPS)
Description: The SHAPS is a 14-item self-report scale to measure hedonic tone. Items (e.g., "I would enjoy reading a book, magazine, or newspaper.") are rated on a 4-point scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree). Either of the 'disagree' responses scores 1 point, and either of the 'agree' responses scores 0 points, for a total scale range of 0-14. Higher scores indicate greater inability to experience pleasure. Patients were asked to rate their experience of the past 24 hours.
Time Frame: as for outcome 3
Population: Several subjects dropped out of the study in between Day 0, Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Day 0 | 7.2222222 (3.9040786) | 7.5500000 (3.9132030) | 6.5909091 (3.2316749) | 7.3500000 (4.1961762) | 6.4736842 (3.7471237)
  Day 1: number analyzed (Participants) | 16 | 19 | 22 | 20 | 18
  Day 1 | 3.9375000 (4.2812576) | 5.7368421 (4.2536534) | 2.22727273 (3.5748036) | 4.3000000 (4.5664682) | 5.0000000 (4.6272848)
  Day 3: number analyzed (Participants) | 15 | 18 | 21 | 20 | 16
  Day 3 | 3.5333333 (3.3777987) | 6.3888889 (4.5262488) | 3.0000000 (3.7815341) | 3.6500000 (4.8370826) | 4.2500000 (3.8384024)
Statistical Analysis 1: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-3.99 to 1.56]
Statistical Analysis 2: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.17, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-1.90 to 3.43]
Statistical Analysis 3: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-5.32 to -0.16]
Statistical Analysis 4: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-3.35 to 1.93]
Statistical Analysis 5: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-3.25 to 2.66]
Statistical Analysis 6: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 6]; Test type: Superiority; p = 0.39, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.76, 95% CI 2-sided [-0.06 to 5.59]
Statistical Analysis 7: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-3.91 to 1.58]
Statistical Analysis 8: Comparison: Ketamine 0.1mg vs Ketamine 0.2mg vs Ketamine 0.5mg vs Ketamine 1.0mg vs Midazolam 0.045mg; [analysis description as in outcome 3, analysis 8]; Test type: Superiority; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-3.22 to 2.35]

8. Secondary Outcome: Clinician-Administered Dissociative States Scale (CADSS) Scores During Infusion
Description: The CADSS is a 23-item self-report scale for the assessment of dissociative states. It is a reliable, valid self-report instrument. The severity of each dissociative symptom ranges from 0 (not present) to 4 (extreme). The total score is calculated by summing across items, with a total possible range of 0-92. The CADSS was administered right before infusion, and 40, 80 minute and 120 minutes after the start of infusion. The timeframe is "at this moment".
Time Frame: Day 0/baseline at 0, 40, 80, and 120 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
units on a scale
  Minute 0 | 0.1111111 (0.4714045) | 0.1000000 (0.4472136) | 0 (0) | 0.1000000 (0.3077935) | 0.4210526 (1.01739326)
  Minute 40 | 3.0000000 (5.0758946) | 4.0500000 (4.2608993) | 14.2727273 (9.6076644) | 24.6842105 (17.7108022) | 2.6842105 (3.5127171)
  Minute 80 | 0.4444444 (0.7838234) | 0.1000000 (0.4472136) | 0.7727273 (2.1141658) | 1.8000000 (2.9664794) | 1.1578947 (1.8337320)
  Minute 120 | 0.0555556 (0.2357023) | 0 (0) | 0.1363636 (0.6396021) | 0.6500000 (1.5985191) | 0.5789474 (0.9015905)

9. Secondary Outcome: Number of Participants Reporting Suicidal Ideation/Behavior on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia Suicide Severity Rating Scale (C-SSRS): The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed in the National Institute of Mental Health Treatment of Adolescent Suicide Attempters Study to assess severity and track suicidal events through any treatment. It is a clinical interview providing a summary of both ideation and behavior that can be administered during any evaluation or risk assessment to identify the level and type of suicidality present. The C-SSRS can also be used during treatment to monitor for clinical worsening or improvement. It contains 5 rating scale questions (yes/no) for suicidal ideation increasing severity and 5 rating scale questions (yes/no) for suicidal behavior of increasing severity. The time frame is for both lifetime and the past six months for the Baseline/Screening scale and since the last visit for the Since Last Visit scale.
Time Frame: Screening Visit and Days 0, 1, 3, 5, 7, 14 and 30 combined
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
Participants
  Screening: # with suicidal ideation/behavior | 17 | 15 | 17 | 14 | 17
  Follow-Up: # with suicidal ideation/behavior | 15 | 9 | 10 | 6 | 13

10. Secondary Outcome: Number of Participants With Abnormal and Clinically Significant CBC and Chemistry Labs by Treatment
Description: 1. CBC
  2. Chemistry (Total bilirubin, AST, ALT, GGT, ALK Phosphatase, Creatinine, BUN/Urea, Glucose, Uric Acid)
  Testing was performed by study site laboratories and used institutional normal lab value ranges.
Time Frame: Day 3 and Early Termination Visit (approximately 3 weeks following intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam 0.045mg
Number analyzed (Participants) | 18 | 20 | 22 | 20 | 19
Participants
  Chemistry ALT(SGPT) | 0 | 1 | 0 | 0 | 0
  Chemistry AST(SGOT) | 0 | 1 | 0 | 0 | 0
  Chemistry Total Bilirubin | 0 | 1 | 0 | 0 | 0
  Chemistry Remaining Tests | 0 | 0 | 0 | 0 | 0
  CBC | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Number of patients with adverse events post infusion (treatment) up to 30 days.
Arm/Group | Ketamine 0.1mg | Ketamine 0.2mg | Ketamine 0.5mg | Ketamine 1.0mg | Midazolam (Active Placebo)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20 | 0/22 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/20 | 0/22 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 17/18 | 18/20 | 14/22 | 17/20 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.1mg (N=18) | Ketamine 0.2mg (N=20) | Ketamine 0.5mg (N=22) | Ketamine 1.0mg (N=20) | Midazolam (Active Placebo) (N=19)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine 0.1mg (N=18) | Ketamine 0.2mg (N=20) | Ketamine 0.5mg (N=22) | Ketamine 1.0mg (N=20) | Midazolam (Active Placebo) (N=19)
Headache (Nervous system disorders) | 3 | 2 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 3 | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Blood Pressure Increase (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Poor Quality Sleep (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Blood Testosterone (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dissociation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (General disorders) | 0 | 0 | 0 | 1 | 0
Exposure to Toxic Agent (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hepatic Enzyme Increased (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Increased Appetite (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Initial Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Intentional Self-Injury (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Malaise (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Overdose (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Presyncope (General disorders) | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Self Injurious Behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vertigo (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
White Blood Cell Count Decreased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No